CLINICAL TRIAL: NCT04334408
Title: A Phase II Double-Blinded Placebo Controlled Individual Subject Stepped Wedge Clinical Trial Evaluating the Safety and Efficacy of Fremanezumab for Migraine in Adult CADASIL
Brief Title: Safety and Efficacy of Fremanezumab for Migraine in Adult CADASIL
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding to support the trial.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James F. Meschia, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18-010786
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Cadasil; Migraine
MeSH Terms: conditions — CADASIL; Migraine Disorders | interventions — fremanezumab; erenumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects with CADASIL treatment intervention (Active Comparator): Subjects that have been diagnosed with both CADASIL and moderately to severely disabling migraine headaches will be treated with Fremanezumab injections.
  Interventions: Drug: Fremanezumab; Drug: Placebo
- Subjects with CADASIL placebo intervention (Placebo Comparator): Subjects that have been diagnosed with both CADASIL and moderately to severely disabling migraine headaches will be treated with placebo injections.
  Interventions: Drug: Fremanezumab; Drug: Placebo

INTERVENTIONS:
Drug: Fremanezumab — Subjects will receive a single dose total 225 mg (1 injection of 225 mg per 1.5 mL injection) followed by a single dose of 225 mg (1 1.5mL injection) at four week intervals. Both the subject and the investigator will be blinded to the timing of transition to and from placebo and the transition to and from fremanezumab.
  Other Names: Ajovy
Drug: Placebo — Placebo injections during the run in and washout serves as the control condition. Both the subject and the investigator will be blinded to the timing of transition to and from placebo and the transition to and from fremanezumab.

SUMMARY:
Researchers are trying to find out more about the side effects of fremanezumab when treating patients with Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy (CADASIL) for migraine headaches.

DETAILED DESCRIPTION:
Subjects will receive 4 to 20 weeks of placebo injections followed by 12 weeks of monthly administered fremanezumab by subcutaneous injection (225 mg split four weeks apart for 12 weeks). Following completion of the 12 weeks of therapy, the participant will return to placebo for the washout period. Both the patient and the investigator will be blinded to the timing of transition to and from placebo and the transition to and from fremanezumab.

ELIGIBILITY:
Inclusion Criteria

* Age 18 to 70 years old
* English speaking
* Diagnosis of CADASIL confirmed by presence of a pathogenic NOTCH3 gene mutation
* Diagnosis of migraine for at least 12 months and diagnosis of chronic migraine for at least 28 days according to the International Classification of Headache Disorders
* MIDAS score of >10 points
* Ability to provide written informed consent

Exclusion Criteria

* History of ischemic stroke within 4 weeks of screening assessment
* Screening blood pressure >150 mm Hg
* Use of onabotulinum toxin A 4 months prior to trial or other injectable/stimulatory/magnetic method of headache control
* Use of opiates or barbiturates 4 days prior to trial
* Patients with competing intracerebral pathology (e.g. history of intracerebral hemorrhage, multiple sclerosis)
* NYHA Class III or IV congestive heart failure
* History of myocardial infarction
* History of coronary bypass surgery or coronary stenting
* Pregnancy or breastfeeding
* Contraindication to undergoing brain MRI per standard clinical practice guidelines
* Vulnerable populations, including incarcerated inmates, dementia, and inability to provide consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in migraine-related disability | Baseline, 2 week intervals up to 48 weeks
  Measured using the The Migraine Disability Assessment (MIDAS) questionnaire which is a brief, self-administered questionnaire designed to quantify headache-related disability over a 3 month period using number of days
Change in headache intensity | Baseline, 2 week intervals up to 48 weeks
  Measured using Headache Impact Test (HIT)-6 scores with the answers being never, rarely, sometimes, very often or always and equating to 6, 8, 10, 11, and 13 points respectively. Each answer is summated to equal the final score.
Adverse events | 48 weeks
  Number of adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: James F Meschia, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials